CLINICAL TRIAL: NCT00010127
Title: A Safety and Feasibility Study of Active Immunotherapy in Patients With Metastatic Prostate Carcinoma Using Autologous Dendritic Cells Pulsed With Antigen Encoded in Amplified Autologous Tumor RNA
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0759; DUMC-000759-00-4R1; DUMC-DORIS-99043; NCI-G00-1910; CDR0000068447 (Other: NCI)
Record Dates: First submitted 2001-02-02; First posted 2003-07-30 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2008-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response to kill prostate tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of autologous dendritic cells transfected with autologous total tumor RNA in patients with metastatic prostate cancer.
* Determine the presence, frequency, and activation status of tumor specific and prostate specific antigen (PSA) specific cellular immune responses in patients treated with this regimen.
* Determine delayed-type hypersensitivity reactions to PSA protein and other recall antigens in patients before and after being treated with this regimen.
* Determine clinical responses based on clinical and biochemical (PSA) response criteria in patients treated with this regimen.
* Determine a platform for immunological treatment using dendritic-cell based tumor vaccines in these patients.

OUTLINE: This is a dose escalation study.

Tumor tissue and peripheral blood stem cells are collected from patients and cultured in vitro with sargramostim (GM-CSF) and interleukin-4 for 7 days to produce dendritic cells (DC). Patients receive autologous DC transfected with autologous prostate carcinoma RNA intradermally once weekly on weeks 0-3 for a total of 4 doses.

Cohorts of 3-6 patients receive escalating doses of DC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at weeks 6, 8, 10, and 12; every 3 months for 9 months; and then annually for 2 years.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the prostate

  * Stage D1-3
  * Regional lymph node, bone, visceral, or soft tissue metastases
  * No transitional cell or small cell carcinoma
* Testosterone less than 50 mg/L if prior treatment with luteinizing hormone releasing hormone (LHRH) analogues or estrogens
* Evidence of androgen refractory disease after surgical castration and discontinuation of LHRH analogue therapy
* No previously irradiated or new CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 6 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* PT at least 11.3 seconds but no greater than 13.3 seconds
* PTT at least 20.1 seconds but no greater than 32.9 seconds
* No hepatic disease
* No viral hepatitis

Renal:

* Creatinine less than 2.5 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* No asthma
* No chronic obstructive pulmonary disease
* No severe lung disease

Other:

* No other medical illness or psychological impediment that would preclude study
* No other concurrent malignancy except nonmelanoma skin cancer or controlled superficial bladder cancer
* No active acute or chronic infection including symptomatic urinary tract infection
* No autoimmune disease (e.g., inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, scleroderma, or multiple sclerosis)
* HIV negative
* Adequate peripheral vein access

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed
* No other concurrent immunotherapy

Chemotherapy:

* Prior chemotherapy allowed
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior non-steroidal hormonal therapy if increase in PSA while receiving non-steroidal hormonal therapy
* At least 6 weeks since prior steroids
* Concurrent LHRH analogues for gonadal androgen suppression allowed
* No concurrent steroid therapy
* No concurrent corticosteroids

Radiotherapy:

* See Disease Characteristics
* Prior palliative radiotherapy for bone metastases allowed
* Prior prostatic radiotherapy allowed
* At least 4 weeks since prior radiotherapy
* At least 12 weeks since prior strontium chloride Sr 89
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior therapy
* No concurrent immunosuppressive agents (e.g., azathioprine or cyclosporine)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2000-11; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Vieweg, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States